CLINICAL TRIAL: NCT02188173
Title: An Observational Study of OZURDEX® in Diabetic Macular Edema (DME)
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: GMA-US-EYE-0272; REINFORCE (Other: Allergan)
Record Dates: First submitted 2014-07-10; First posted 2014-07-11 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Macular Edema
MeSH Terms: conditions — Macular Edema | interventions — Calcium Dobesilate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- dexamethasone 700 ㎍ intravitreal implant: Patients who receive dexamethasone 700 ㎍ (OZURDEX®) intravitreal implant treatment for Diabetic Macular Edema. All decisions regarding treatment are made at the sole discretion of the treating physician in accordance with their usual practices.
  Interventions: Drug: dexamethasone 700 ㎍ intravitreal implant

INTERVENTIONS:
Drug: dexamethasone 700 ㎍ intravitreal implant — Patients who receive dexamethasone 700 ㎍ (OZURDEX®) intravitreal implant treatment for Diabetic Macular Edema. All decisions regarding treatment are made at the sole discretion of the treating physician in accordance with their usual practices.
  Other Names: OZURDEX®

SUMMARY:
This is a study of OZURDEX® use in clinical practice in patients with diabetic macular edema (DME).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DME in at least one eye treated OZURDEX® per clinical practice

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetic macular edema (DME) treated with (OZURDEX®) in clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Maximum Change from Baseline in Best Corrected Visual Acuity (BCVA) in the Study Eye | Baseline, 12 Months
Percentage of Patients with a BCVA Improvement of ≥15 Letters in the Study Eye | Baseline, 12 Months
Average Change from Baseline in BCVA in the Study Eye | Baseline, 12 Months

SECONDARY OUTCOMES:
Percentage of Patients with an Increase from Baseline of ≥2 Lines in BCVA in the Study Eye | Baseline, 12 Months
Percentage of Patients with an Increase from Baseline of ≥3 Lines in BCVA in the Study Eye | Baseline, 12 Months
Percentage of Patients with BCVA of 20/40 or Better in the Study Eye | Baseline, 12 Months
Mean Number of Ozurdex Injections in the Study Eye | 12 Months
Mean Time Between Ozurdex Injections in the Study Eye | 12 Months
Change from Baseline in Central Retinal Subfield Thickness (CRT) in the Study Eye | Baseline, 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (18):
- United States (18):
  - Retinal Consultants of Phoenix, Phoenix, Arizona
  - West Coast Retina, San Francisco, California
  - Orange Co Retina Medical Group, Santa Ana, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Colorado Retina Associates, Denver, Colorado
  - Illinois Retina Associates, Harvey, Illinois
  - Raj Maturi, MD PC, Indianapolis, Indiana
  - John-Kenyon American Eye Institute, New Albany, Indiana
  - Associated Retina Consultants, Royal Oak, Michigan
  - Associated Retinal Consultants, PC, Traverse City, Michigan
  - Lifelong Vision Foundation, Chesterfield, Missouri
  - Eyesight Ophthalmic Services, Portsmouth, New Hampshire
  - New Jersey Retina, New Brunswick, New Jersey
  - Long Island Vitreoretinal Consultants - Long Island Retina - Hauppauge, Great Neck, New York
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Texas Retina Associates, Arlington, Arlington, Texas
  - Valley Retina Institute, P.A., McAllen, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas